CLINICAL TRIAL: NCT02379702
Title: Turkey Metabolic Syndrome Prevalence Study - METSAR II
Brief Title: Metabolic Syndrome Prevalence Study
Status: Completed | Type: Observational
Sponsor: Abdi Ibrahim Ilac San. ve Tic A.S. (Industry)
Responsible Party: Sponsor
Other Study IDs: METSAR-II
Record Dates: First submitted 2014-10-17; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — ANAPC16 protein, human

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Metabolic Syndrome — This study will provide important information on the social and economic dimensions of metabolic syndrome

SUMMARY:
Following the first study conducted to investigate the prevalence of metabolic syndrome and its components in Turkey, it was aimed to demonstrate the change in general health condition of available patients after the period of time lapsed. This study will provide important information on the social and economic dimensions of metabolic syndrome and will contribute to development of preventive programs.

DETAILED DESCRIPTION:
In the first METSAR-I study conducted in 2003, metabolic syndrome screening was made by two different team. Participants were visited at their addresses and informed about the research study and gave written consent. They were invited on an empty stomach for hospital visit on the day after. Pre-trained nurses completed the forms of patients during that second visit. After 11 years, a questionnaire by telephone survey will be applied to patients who participated in the METSAR-II study. The main goal is to determine the changes of metabolic syndrome population during that period.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who participated in the METSAR-I study in 2003
* Patients who accepted to participate will be included the second follow up phase.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The previous study included 4.264 patients from 47 cities and we are going to try to get in contact all those patients. Data obtained from available patients will be analysed and the change trend will be evaluated
Sampling Method: Non-Probability Sample
Enrollment: 1659 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
comorbidities and changes in general health | 10 year

CONTACTS AND LOCATIONS:
Overall Officials: Omer Kozan, Study Director — Dokuz Eylul University
Locations (6):
- Turkey (Türkiye) (6):
  - Ankara University, Ankara
  - Gazi University, Ankara
  - Yuksek Ihtisas Hospital, Ankara
  - Istanbul Cerrahpasa University, Istanbul
  - Istanbul Medeniyet University, Istanbul
  - Prof. Dr. Omer Kozan, Izmir